CLINICAL TRIAL: NCT07047105
Title: Investigation of the Acute Effects of Nepalese Pepper Extract (Zanthoxylum Armatum DC) on Cognitive Function, Mood and Gaming Performance in Young, Healthy, Competitive Gamers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Mibelle Group Biochemistry (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 53BS2
Record Dates: First submitted 2025-06-04; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cognition; Mood; Gaming Performance; Fatigue
Keywords: Cognition; Mood; Gaming; Performance; Esports; Nepalese Pepper; Timut Pepper; Zanthoxylum Armatum; Fatigue
MeSH Terms: conditions — Fatigue | interventions — Caffeine

STUDY DESIGN:
Intervention Model Description: Randomised, double-blind, placebo-controlled, four-arm crossover design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Treatment will be blinded according to the randomisation schedule by a researcher who has no other involvement in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ZA 150mg (Experimental): 150mg dosage of Nepalese Pepper (Zanthoxylum Armatum) extract in capsule form. Consumed during testing visit to measure acute effects over day of consumption.
  Interventions: Dietary Supplement: Nepalese Pepper (Zanthoxylum Armatum) extract 150mg
- ZA 300mg (Experimental): 300mg dosage of Nepalese Pepper (Zanthoxylum Armatum) extract in capsule form. Consumed during testing visit to measure acute effects over day of consumption.
  Interventions: Dietary Supplement: Nepalese Pepper (Zanthoxylum Armatum) extract 300mg
- Caffeine (Active Comparator): 75mg dose of caffeine (Caffeine anhydrous Pulver) in capsule form. Consumed during testing visit to measure acute effects over day of consumption.
  Interventions: Dietary Supplement: Caffeine 75mg
- Placebo (Placebo Comparator): Inert placebo, Microcristalline Cellulose MCC, delivered in capsule in form.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nepalese Pepper (Zanthoxylum Armatum) extract 150mg — The intervention is a powdered form of Zanthoxylum Armatum (ZA) extract delivered in capsule form. The dosage is 150mg.
  Other Names: Timut Pepper
  Arms: ZA 150mg
Dietary Supplement: Nepalese Pepper (Zanthoxylum Armatum) extract 300mg — The intervention is a powdered form of Zanthoxylum Armatum (ZA) extract delivered in capsule form. The dosage is 300mg.
  Arms: ZA 300mg
Dietary Supplement: Placebo — Microcristalline Cellulose MCC
  Arms: Placebo
Dietary Supplement: Caffeine 75mg — Caffeine anhydrous Pulver, 75mg
  Arms: Caffeine

SUMMARY:
The goal of this clinical trial is to learn if a Nepalese Pepper Extract (Zanthoxlum Armatum, ZA) supplement can improve cognitive performance and mental abilities in competitive gamers aged 16 to 34. The main questions it aims to answer are:

1. Does ZA supplement improve cognitive abilities like attention, memory, and decision-making?
2. What is the most effective dose of ZA supplement (300mg vs 150mg)?
3. How do the effects of ZA supplement compare to caffeine?

Researchers will compare four different treatments (high-dose ZA, low-dose ZA, caffeine, and placebo) to see if ZA supplement produces better cognitive performance than placebo and how it compares to caffeine**.

Participants will:

* Complete a screening visit with health checks and training on computer tasks
* Attend four testing visits (7-14 days apart) where they receive different treatments
* Avoid alcohol and energy drinks for 24 hours before each visit, and caffeine from waking
* Take assigned treatment at 11:30am and complete cognitive tests at -1, 1, 3, and 5 hours in relation to dose.
* Complete mood questionnaires, sleep assessments, and gaming-specific tasks (aim training, character control)
* Wear heart rate monitors during testing
* Eat standardized meals provided during visits
* Play competitive games at home in the evening and complete performance questionnaires

DETAILED DESCRIPTION:
Zanthoxylum armatum DC (ZA), also known as Nepalese pepper (or TImut pepper, contains numerous active chemicals throughout all parts of the organism. Traditionally used in the treatment of intestinal disorders, depression and as topical treatment for toothache it is commonly ingested through the form of Daikenchuto, a traditional combination of the Zanthoxylum fruit with ginseng root, ginger rhizome and rice gluten. In recent years it has been established that ZA also possesses cognitive enhancing properties, with the primary active component revealed to be the fatty acid amide hydroxy α-sanshool. Additionally, ZA is rich in monoterpenes which have also been shown to positively affect cognition and the combination of these compounds may lead to numerous improvements in brain function.

Through a double-blind placebo-controlled study, acute single dose administration of 80 mg of ZA was shown to improve cognitive performance in 'Speed of Attention' and Rapid Visual Information Processing, a sustained attention task. In the same study, chronic (56 day) administration resulted in overall improvement in 'Speed of Performance' with more correct Serial 3 subtractions 3h post dose and lower mental fatigue compared to placebo during performance of the Cognitive Demand Battery (CDB). In both acute and chronic cases, the mechanisms underpinning the effects are currently unknown, and the differences could be attributed to distinct changes over time. For the acute effects there may be a cholinergic mechanism at play, with previous research suggesting that there has been a cholinesterase inhibitory effect from ZA. Meanwhile, the observed chronic improvements suggest a more general improvement in neural efficiency and processing speeds rather than the memory/attention benefits generally expected from cholinergic agents. A similar study on the cognitive effects of a multi-ingredient herbal supplement also resulted in speed of cognition improvement. Although this herbal remedy did not contain ZA or hydroxy α-sanshool, it did contain short chain fatty acids and terpenes suggesting a similar mechanism could be at work to improve neural efficiency.

An increasing area of interest for performance research is in the world of Esports and competitive gaming, where cognitive abilities are paramount. As with non-digital sports, esport competition incurs physical and mental demands, including motor skills, mental agility, processing speed, motivation, executive function and to a lower degree, physical exertion. Success hinges on mastering cognitive tasks such as visuospatial processing, cognitive workload, attention and cognitive control, hand-eye coordination, fast reaction times and quick decision-making capabilities. Alongside these cognitive factors, the importance of personal social and emotional competencies within esports has been explored through the creation of a detailed competence model of digital games. Factors such as self-efficacy, mood, self-control, personality traits and emotional self-regulation have displayed correlations with traditional sport performance and therefore it would be expected improvements in these areas would also create better results for gamers. Within esports, viewership is overwhelmingly dominated by either Massive Online Battle Arena's (MOBA) and First Person Shooters (FPS), according to peak viewing statistics in recent years. It has been noted that FPS and MOBA game types share a similar fast paced, high intensity element which separates them from Real-time Strategy (RTS) games, however despite this the contrast in player character control mechanisms creates distinct performance metrics. Consequently, studies looking to analyse game performance across different genre players should incorporate genre-specific game performance measurement tools, the simplest of which would be in-game rank, but could extend to more detailed in-game metrics.

Cognitive tests provide a useful measure of the varying domains of mental performance, with a long-established history of validated measures of perception, attention and concentration, memory, executive function and processing speed. Given their broad range of applicability, measures of cognition may be able to map onto varying game genre competencies, as has been seen through research on numeric ability and flexible thinking, establishing some general abilities that persist across all game genres as fundamental cognitive abilities for performance.

One aspect common to all esports players is the prolonged nature of training and gameplay, requiring sustained attention, resulting in high mental demand and fatigue. Energy drink consumption is high within gamers; marketing of these products includes claims of mental fatigue attenuation and maintaining alertness during game play and several energy drink companies also provide sponsorship for esports teams. An emerging area of research considers the potential to enhance gaming performance following administration of various nootropics, primarily focussing on highly caffeinated energy products. Notably here, following 3 mg/kg caffeine, professional gamers performed quicker during a simple reaction time task, alongside quicker and more accurate performance on a first-person shooting task. Similarly, following acute supplementation with 125 mg caffeine, participants were more accurate during a tracking task. Within the same trial, following a combined supplement of caffeine, methylliberine and theacrine (125, 75 and 50 mg, respectively), improvements were observed in visuospatial working memory, alongside quicker kill time within a first-person shooter game and improved self-assessed performance, suggesting a potential synergistic effect when co-supplementing, rather than administering caffeine in isolation. A second trial using the same combined supplement that focused on traditional cognitive test outcomes reported improved performance on the Flanker Test of Inhibitory Control and quicker reaction time on the Psychomotor Vigilance Task; alongside increased self-reported alertness.

The high caffeine content in these products is, however, linked to several undesirable side effects, including heightened jitteriness and tension, as well as decreased deep sleep and overall sleep duration. These effects can negatively impact both short-term and long-term gaming performance. As gaming becomes a more viable career, gamers are likely to become more aware of these negative effects and seek healthier alternatives. This has sparked interest in finding non-caffeinated options to combat mental fatigue and enhance gaming performance. A previous trial assessed the effects of an inositol-enhanced arginine silicate supplement on cognitive and gaming performance. While video game performance remained unchanged, the supplement improved cognitive performance, with quicker completion time and fewer errors on the Trail Making Test, improved performance on the Stroop task and increased self-reported vigour. These findings suggest improvements in executive functioning, processing speed, task switching, and selective attention, suggesting the potential for game-related improvements to cognitive function from non-caffeinated supplements.

The previous intervention study conducted by our group administered 2.8 g Zanthoxylum armatum DC. medium-chain triglyceride (MCT) oil extract (corresponding to 80 mg Z.armatum DC.). Each 2.8 g dose contained alkamides including 7.8 mg hydroxy α-sanshool and monoterpenes including 5.3 mg limonene, 3.6 mg linalool and 2.3 mg methyl cinnamate. A new formulation of ZA delivered through a powder rather than a liquid format will be used in the proposed study, allowing for varying dosage amounts to be tested to ascertain the effects of ZA at lower doses. The main aim of the current study is therefore to investigate the acute cognitive and mood effects of ZA in young, healthy competitive gamers. A focused acute study with a crossover design may lead to more in depth coverage of the attention changes in cognitive abilities under acute doses of ZA, while also providing an opportunity to reveal if overall neural efficacy can be observed at this level. Additional aims include: discovering if lower dosages of the supplement than previously used in research are effective; ascertaining if cognitive improvements translate to objective and subjective in-game performance improvements in different genre players; to deepen understanding of how different genres of Esport present different cognitive gameplay requirements and investigate how differing genre players can be assessed within a single study.

Primary objectives

The primary objectives of this study are to evaluate the acute effects of 150 and 300 mg of the powdered formulation of ZA within a young healthy population, with focus on:

* 'Speed of Attention' (RVIP, SRT and CRT)
* Subjective fatigue (CDB)

These were the areas of improvement ascertained by Kennedy et al. (2019) and these results will be tested for replicability. In order to fulfil these objectives, participants will be tested using computerised cognitive tasks (COMPASS) and an online questionnaire in a crossover design, with pre-dose, 1hr post-dose, 3hr post-dose and 5hr post-dose.

Secondary objectives The secondary objectives of this study are to evaluate other cognitive areas where no significant changes were revealed in the previous study, to test for replication and see if any other changes appear. These include

* Accuracy of Attention (RVIP and CRT)
* Speed of Performance (Numeric Working Memory, SRT, CRT, RVIP, Stroop, Delayed Picture Recognition, Delayed Word Recognition)
* Accuracy of Performance (Immediate Word Recall, CRT, Corsi Blocks, RVIP, Stroop, Delayed Word Recall, Delayed Picture Recognition, Delayed Word Recognition)
* Working memory (Numeric Working Memory, Corsi Blocks)
* Speed of memory (Numeric Working Memory, Delayed Picture Recognition, Delayed Word Recognition)
* Episodic memory (Immediate Word Recall, Delayed Word Recall, Delayed Picture Recognition, Delayed Word Recognition)
* Executive Function (Peg and Ball, Stoop interference)

To fulfil these objectives, the full battery of COMPASS tasks will be tested pre-dose, 1hr post-dose, 3hr post-dose and 5hr post-dose, under four differing treatment groups.

In addition, subjective alertness and mental fatigue will also be assessed following each of 3 completions of the Cognitive Demand Battery (CDB). The objective of this battery is to assess the impact of the intervention on speed/accuracy and mental fatigue during continuous performance of cognitively demanding tasks. Participants complete the 10-minute battery of tasks three times in immediate succession (i.e. for a continuous period of 30 minutes). Application of this battery has been shown to reliably increase self-ratings of 'mental fatigue' and to be sensitive to a number of herbal and natural interventions (Kennedy et al., 2008a; D. O. Kennedy & A. B. Scholey, 2004; Reay et al., 2005; Reay et al., 2006).

In addition to this, mood and sleep will also be recorded on testing visits through:

* Positive and Negative Affect Schedule (PANAS)
* Visual Analogue Mood Scales (VAMS)
* Sleep disturbance short form (PROMIS) Heart Rate Variability will also be assessed during select portions of the testing to ascertain if any change in this metric can be matched with either cognitive or gameplay improvements and the treatments.

Further secondary objectives are to implement gaming and gaming-like tasks to assess if any differences can be observed in gameplay related outcomes following treatments. These will include:

* Aim trainer (an aiming game which will challenge the participants to complete mouse accuracy tasks mimicking First Person Shooter (FPS) gameplay)
* Massive Online Battle Arena (MOBA) control simulator (a game/training simulation using the controls and perspective of MOBA games to test movement and input ability)
* Multi-Tasking Framework (MTF)
* Finger Tapping Task (FTT)

In addition to this, gameplay monitoring of at home play will be implemented to provide a basis for assessment of gameplay ability in a further chronic study. These measures are exploratory and they may not be analysed if compliance with at home gaming requests is inconsistent. This will include:

* Subjective Performance Gameplay Scale (for participants to complete at home after playing a competitive video game on the evening of their treatment day)
* Gameplay tracking (tracking of games played by participants to view the quality of their performances on the evening of the treatment day) These additional measures of gameplay performance will be assessed with the intention of building a robust method of assessing gameplay performance over a longer period.

INVESTIGATIONAL PLAN Trial Design and Plan This study will follow a randomised, placebo-controlled, double-blind, crossover design. Participants will attend the lab on five separate occasions which will include a screening/training visit and four testing visits under each of the treatments within the protocol.

Trial population A total sample of 60 participants will take part in this study. Criteria will be checked at screening and continued adherence to them will be checked during the pre-test interview on each visit.

Following informed consent eligible participants will undergo training on the computerised cognitive tasks and gaming tasks. The training session will follow standard operating procedures to decrease the chance of learning effects during the main trials.

Testing Visits 1, 2, 3 and 4 (7+/-3 days between each visit)

Participants will be asked to avoid alcohol and refrain from intake of 'over the counter' medication for 24 hours. The participants will also be asked to refrain from consuming energy drinks for 24 hours prior to their testing visit, and to not consume caffeine from waking before each testing visit. Participants will be contacted to remind them of the requirements prior to each visit. On the morning of Testing Visit 1, participants will be requested to eat a simple breakfast of plain cereal and milk or toast and butter at least 1 hour prior to arrival at the laboratory (also avoiding any caffeinated products); the time and composition of breakfast will be standardised across all visits. During their testing visits, the participants will be asked to avoid consumption of any other food or liquids aside from water and the lunch and snacks provided by the research team. Participants will report to the Brain, Performance and Nutrition Research Centre at Northumbria University between 9:45am and 10 am for each visit. The following procedures will be required before commencement of the trial:

* Review continued conformity with the inclusion and exclusion criteria
* Adverse event assessment
* Assessment that participant is not unwell and is well-rested
* Randomisation of participant (Visit 1 only)

At 10:10am gaming tasks will be performed by the participants. Following this at 10:30am the first round of cognitive tests will begin for 1 hour. At the end of this round of tests the treatments will be administered, with each participant receiving a random treatment in accordance with the randomisation schedule.

Figure 1. Day schedule of participant's testing visits. Following treatment, a 40 minute break will take place, followed by gaming tasks for 20 minutes and then at 12:30pm the second round of cognitive tests (1hr post-dose) will occur. Before each round of cognitive tests 20 minutes of gaming related tasks will be performed. After these cognitive tests lasting around 1 hour, a standardised lunch will be provided, consisting of a cheese sandwich, ready salted crisps, and a custard pot, around 1:30 pm. Additionally, they will be offered an optional snack of digestive biscuits following the 3hr post-dose assessment at approximately 3:30 pm. The final round of cognitive tests will start at around 4:30pm with the testing day ending at 5:30pm.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 to 34 years inclusive
* Males and females
* Self-report of good health
* Usually a regular (at least once per week) player of competitive multiplayer games, (prospective participants will be asked to contact the researchers to discuss their gaming habits if uncertain that they meet the criteria).

Exclusion Criteria:

* Have any pre-existing medical condition/illness which will impact taking part in the study (i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance).
* Are currently taking prescription medications NOTE: the explicit exceptions to this are contraceptive treatments for female participants, and those taken 'as needed' in the treatment of asthma and hay fever. There may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening.
* Have high blood pressure (systolic over 139 mm Hg or diastolic over 89 mm Hg); or have low blood pressure (systolic below 90 mm Hg or diastolic below 60 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2
* Are pregnant, seeking to become pregnant or lactating
* Have learning and/or behavioural diagnoses such as dyslexia or ADHD
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products
* Excessive caffeine intake (> 500 mg per day). If participants consume energy drinks they will be asked to refrain from this for 24 hour prior to attending testing.
* Have relevant food intolerances/sensitivities, including caffeine sensitivity.
* Have taken antibiotics within the past 4 weeks
* Have taken dietary supplements e.g. Vitamins, omega 3 fish oils etc. in the last 4 weeks (Note: participation is possible following a 4-week supplement washout prior to participating and for the duration of the study on the proviso that the supplements they are taken are out of choice and not medically prescribed or advised)
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have done so in the past 4 weeks
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disorders or are taking sleep aid medication
* Any known active infections
* Are non-compliant with regards treatment consumption

Ages: 16 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Speed of Attention | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through performance on Rapid Visual Information Processing, Simple Reaction Time and Choice Reaction Time
Subjective Fatigue | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Following completion of Cognitive Demand Battery subjective fatigue will be assessed through self assessment of fatigue levels.

SECONDARY OUTCOMES:
Accuracy of Attention | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through combined performance on Rapid Visual Information Processing and Choice Reaction Time tasks
Speed of Performance | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through combined performance on Numeric Working Memory, SRT, CRT, RVIP, Stroop, Delayed Picture Recognition, Delayed Word Recognition
Accuracy of Performance | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through combined performance on Immediate Word Recall, CRT, Corsi Blocks, RVIP, Stroop, Delayed Word Recall, Delayed Picture Recognition, Delayed Word Recognition
Working memory | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through combined performance on Numeric Working Memory, Corsi Blocks
Speed of memory | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through combined performance on Numeric Working Memory, Delayed Picture Recognition, Delayed Word Recognition
Episodic memory | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through combined performance on Immediate Word Recall, Delayed Word Recall, Delayed Picture Recognition, Delayed Word Recognition
Executive Function | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Score calculated through score on Peg and Ball and Stroop interference
Mood | Prior to intervention on each testing visit for each arm, along with post dose 1 hour, post dose 3 hour and post dose 5 hour.
  Mood rating calculated through answers to Visual Analogue Mood Scales and Positive and Negative Affect Schedule
Heart Rate Variability (HRV) | Prior to intervention on each testing visit for each arm, along with post dose 40 minutes, post dose 160 minutes and post dose 220 minutes.
  HRV
Multi Tasking Ability | Prior to intervention on each testing visit for each arm, along with post dose 40 minutes, post dose 160 minutes and post dose 220 minutes.
  Multi Tasking Ability measured through Multi Tasking Framework score
First Person Shooter Aiming Ability | Prior to intervention on each testing visit for each arm, along with post dose 40 minutes, post dose 160 minutes and post dose 220 minutes.
  First Person Shooter Aiming Ability with a mouse measured through performance on an aim trainer (Aim Labs)
Finger Tapping Task | Prior to intervention on each testing visit for each arm, along with post dose 40 minutes, post dose 160 minutes and post dose 220 minutes.
  Number of finger taps in 10 seconds
MOBA Control Ability | Prior to intervention on each testing visit for each arm, along with post dose 40 minutes, post dose 160 minutes and post dose 220 minutes.
  Measure of character control ability using a custom MOBA style game to test movement and input ability.
Subjective Gameplay Performance | At home on the evening at least 6 hours post dose, on each testing visit following gameplay.
  Subjective Performance Gameplay Scale self report by participants
Tracked Game Performance | At home on the evening at least 6 hours post dose, on each testing visit following gameplay.
  Online tracking of game performance using participant game profile information to assess performance through various in game metrics.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University - Brain Performance and Nutrition Research Centre, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: No